CLINICAL TRIAL: NCT01729052
Title: The Effect of Acupuncture for Alleviation of Postoperative Nausea, Vomiting, and Pain in Children: The Implications of Parental Attitudes and Expectations
Brief Title: Acupuncture for Postoperative Nausea, Vomiting and Pain in Children: The Implication of Parental Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012/631
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Postoperative Nausea and Vomiting; Postoperative Pain
Keywords: Acupuncture; Children; Postoperative nausea and vomiting; Postoperative pain; Parental attitudes; Parental expectations
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture and standard treatment (Experimental): Acupuncture at Neiguan (Pericardium-6) bilaterally with Seirin needles no 3 (0.20x15 mm) to a depth of approximately 7 mm will be performed on the children immediately after induction of anaesthesia and removed before they are fully awake.
  Standard treatment: general anaesthesia
  Interventions: Device: Acupuncture
- Standard treatment (No Intervention): General anaesthesia

INTERVENTIONS:
Device: Acupuncture
  Arms: Acupuncture and standard treatment

SUMMARY:
Postoperative nausea and vomiting (PONV) remain a significant challenge in our practice. However, pharmaceutical prophylaxis is only partially effective and can imply unpleasant adverse effects. Accordingly, the use of non-pharmacological methods in preventing PONV is appropriate. Acupuncture is reported to reduce PONV and pain, and the adverse events are minimal.

The objective of this multicentre, double-blinded, randomized, controlled trial is to investigate whether acupuncture can be a supplementary to the ordinary treatment in children undergoing tonsillectomy and/or adenoidectomy. In addition, the non-specific effect of parental attitudes and expectations on the outcomes will be explored.

Two hundred and eighty patients will be included and randomized into two groups

1. Treatment group: acupuncture treatment (approximately 15 to 20 minutes) during anaesthesia and standard treatment
2. Control group: standard treatment

The primary endpoints in the intervention study are nausea, retching, vomiting and pain during 24 hours postoperatively. The effect of acupuncture will be studied with regard to any association with possible factors of predisposition to PONV, as well as with other factors registered during the study. Adverse events from acupuncture will be registered.

The objective of the self-report questionnaires is to

* investigate parental attitudes and expectations to the acupuncture treatment pre- and postoperatively
* compare data of the outcomes from the intervention trial with data from the questionnaires, in order to find any correlation between parental beliefs, attitudes and expectations, and the effect of the acupuncture treatment

ELIGIBILITY:
Inclusion Criteria:

* Children from two to eleven years of age
* Children scheduled for tonsillectomy and/or adenoidectomy
* Informed consent from the parents

Exclusion Criteria:

* American Society of Anesthesiologists grade greater than or equal to III (patient with severe systemic disease)
* Patients/parents in need of an interpreter
* Rash or local infection over an acupuncture point
* Emesis during the previous 24 hours
* Use of medication with antiemetic effect within the 24 hours before surgery
* Gastric or intestinal diseases

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea Postoperative vomiting Postoperative pain | Within 24 hours postoperatively

OTHER OUTCOMES:
Parental attitudes Parental expectations | Within 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Arne Johan Norheim, dr.phil., Principal Investigator — NAFKAM, UiT

REFERENCES:
- [Derived] Liodden I, Pripp AH, Norheim AJ. Placebo by proxy expectations toward acupuncture change over time: a survey comparing parental expectations to acupuncture pre- and postoperatively. BMC Complement Altern Med. 2018 Jun 14;18(1):183. doi: 10.1186/s12906-018-2248-z. PMID 29898710
- [Derived] Liodden I, Sandvik L, Norheim AJ. Placebo by Proxy--the Influence of Parental Anxiety and Expectancy on Postoperative Morbidities in Children. Forsch Komplementmed. 2015;22(6):381-7. doi: 10.1159/000442565. Epub 2015 Dec 7. PMID 26840420
- [Derived] Liodden I, Sandvik L, Valeberg BT, Borud E, Norheim AJ. Acupuncture versus usual care for postoperative nausea and vomiting in children after tonsillectomy/adenoidectomy: a pragmatic, multicentre, double-blinded, randomised trial. Acupunct Med. 2015 Jun;33(3):196-203. doi: 10.1136/acupmed-2014-010738. Epub 2015 Apr 13. PMID 25870177